CLINICAL TRIAL: NCT03073499
Title: A Single-centre, Non-randomized, Prospective, Open Clinical Trial to Evaluate the Sensitivity of a Number of Clinical and Psychological Outcome Measures for Cancer Patients Being Treated at the Hospital Day Care Unit or (Partially) at Home
Brief Title: A Clinical Trial to Evaluate the Sensitivity of a Number of Clinical and Psychological Outcome Measures for Cancer Patients Being Treated at the Hospital Day Care Unit or (Partially) at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital Groeninge (Other)
Responsible Party: Principal Investigator, Koen Van Eygen, Dr, General Hospital Groeninge
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GHGroeninge
Record Dates: First submitted 2017-02-07; First posted 2017-03-08 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): (Partial) Oncological Home Hospitalization
  Interventions: Procedure: Oncological Home Hospitalization
- Control (No Intervention): Standard oncological treatment at the hospital day care unit

INTERVENTIONS:
Procedure: Oncological Home Hospitalization
  Arms: Intervention

SUMMARY:
This pilot study aims to evaluate the sensitivity, variability and responsiveness of a number of predefined clinical and psychological outcome measuring tools in an ambulant cancer treatment setting (home vs. hospital). The measuring tools will be evaluated in two patient cohorts. One cohort is treated as per standard of care at the outpatient hospital, the other cohort is receiving (partial) cancer treatment at home. A second objective is to create a costs inventory representing total costs for an ambulant treated cancer patient.

ELIGIBILITY:
Inclusion Criteria:

* Starting new oncological treatment at the outpatient hospital.
* ECOG ≤ 2
* Living within 30 minutes of drive from the hospital

Exclusion Criteria:

* Important comorbidity (ECOG > 2)
* Simultaneous radiotherapy treatment
* Language barriers or communication difficulties
* Problematic venous access
* Known problems with administration of the therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the questionnaires FACT-G, EQ-5D and MYCaW to measure quality of life in patients being treated at different ambulatory care settings (hospital vs home) | 8 weeks
  Sensitivity will be analysed by comparing average outcome-scores between both groups
Sensitivity of the questionnaire OUT-PATSAT35 to measure satisfaction with the provided care of patients being treated at different ambulatory care settings (hospital vs home) | 8 weeks
  Sensitivity will be analysed by comparing average outcome-scores between
Sensitivity of the questionnaire HADS to measure anxiety and depression in patients being treated at different ambulatory care settings (hospital vs home) | 8 weeks
  Sensitivity will be analysed by comparing average outcome-scores between outcome responses within both groups
Sensitivity of the questionnaire Distress Barometer to measure distress in patients being treated at different ambulatory care settings (hospital vs home) | 8 weeks
  Sensitivity will be analysed by comparing average outcome-scores between outcome responses within both groups
Sensitivity of a self-designed questionnaire to measure the safety feeling of patients being treated at different ambulatory care settings (hospital vs home) | 8 weeks
  Sensitivity will be analysed by comparing average outcome-scores between outcome responses within both groups

SECONDARY OUTCOMES:
Costs inventory representing total costs for an ambulant treated cancer patient | 8 weeks
  Patients will be asked to record their medical consumptions during the first 8 weeks of treatment using a costs form. Furthermore, also hospital financial data wil be implemented in the costs inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Koen Van Eygen, MD, Principal Investigator — General Hospital Groeninge
Locations (1):
- GH Groeninge, Kortrijk, West Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cool L, Missiaen J, Vandijck D, Lefebvre T, Lycke M, De Jonghe PJ, Vergauwe P, Foulon V, Pottel H, Debruyne P, Van Eygen K. An observational pilot study to evaluate the feasibility and quality of oncological home-hospitalization. Eur J Oncol Nurs. 2019 Jun;40:44-52. doi: 10.1016/j.ejon.2019.03.003. Epub 2019 Mar 23. PMID 31229206